CLINICAL TRIAL: NCT04984382
Title: Comparison of the Effect of Helicobacter Pylori Eradication Before and After the Training of Gastroenterologists on Standardized Helicobacter Pylori Eradication Therapy
Brief Title: Comparison of the Effect of Helicobacter Pylori Eradication Before and After the Training of Gastroenterologists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, doctoral supervisor of Qilu Hospital gastroenterology department, Shandong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021SDU-QILU-G004
Record Dates: First submitted 2021-07-27; First posted 2021-07-30 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Standardized training on Helicobacter pylori eradication; Gastroenterologist

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- After receiving standardized training on Helicobacter pylori eradication (Experimental): After the gastroenterologists receive standardized training to eradicate Helicobacter pylori, they recruit Helicobacter pylori-positive patients for treatment.
  Interventions: Behavioral: Standardized training on Helicobacter pylori eradication treatment
- Before receiving standardized training on Helicobacter pylori eradication (No Intervention): Gastroenterologists recruited patients with Helicobacter pylori positive for treatment before receiving standardized training on Helicobacter pylori eradication.

INTERVENTIONS:
Behavioral: Standardized training on Helicobacter pylori eradication treatment — Standardized training on Helicobacter pylori eradication treatment
  Arms: After receiving standardized training on Helicobacter pylori eradication

SUMMARY:
The researchers recruited gastroenterologists. Physician subjects recruited Helicobacter pylori-positive patients before and after receiving standardized training on Helicobacter pylori eradication. There are no restrictions on treatment options and drugs during the trial. Compare the eradication rate, adverse reaction rate, and patient compliance before and after physician training.

DETAILED DESCRIPTION:
The researchers recruited gastroenterologists to participate in the study, and gastroenterologists recruited Helicobacter pylori-positive patients. In this process, the patient population is not limited, and the eradication program is not limited. Gastroenterologists can follow up or not follow up according to their original diagnosis and treatment. Researchers follow up and record the patient's medication status and adverse reactions in the medication process by phone or WeChat, and evaluate patient compliance. Record the eradication rate. After waiting for all patients admitted by gastroenterologists to be eradicated and re-examined, we will provide standardized Helicobacter pylori eradication training for gastroenterologist subjects. After the training, gastroenterologists recruit Helicobacter pylori-positive patients here. In this process, the patient population is not limited, and the eradication program is not limited. Gastroenterologists can follow up or not follow up according to their original diagnosis and treatment. Researchers follow up and record the patient's medication status and adverse reactions in the medication process by phone or WeChat, and evaluate patient compliance. Record the eradication rate. Compare the eradication rate, the incidence of adverse reactions, and the compliance of the patients before and after the training of the gastroenterologists.

ELIGIBILITY:
Inclusion Criteria:

* 1.Physician specialized in gastroenterology.
* 2.Diagnosis and treatment conditions for H. pylori exist in the hospital where the gastroenterology doctor is located.

(C13 urea breath test, C14 urea breath test, rapid urease test, stool H. pylori antigen test, histopathological test, H. pylori culture, any of the above)

Exclusion Criteria:

* 1.Those who are unable or unwilling to provide informed consent.
* 2.Patients with H. pylori have never been diagnosed and treated.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 1 year
  The eradication rate of before and after the gastroenterologists receiving standardized Helicobacter pylori eradication training

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Xiuli Zuo, Jinan, Shandong, China